CLINICAL TRIAL: NCT07182461
Title: The Effects of Blood Flow Restriction-based Abdominal draw-in Maneuver on Activation of Abdominal Core Muscles in Patients With Non-specific Low Back Pain
Brief Title: The Effects of Dynamic Taping Combined With Corrective Exercises on Cervical Proprioception and Muscle Imbalance in Patients With Upper Crossed Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH113-REC3-197
Record Dates: First submitted 2025-06-11; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Upper Crossed Syndrome
Keywords: posture; muscle imbalance; proprioception
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Combined Dynamic Taping and Corrective Exercise (DT+EX Group) (Experimental): Participants in this group received postural taping using dynamic tape aimed at correcting forward head posture, rounded shoulders, and thoracic kyphosis. The tape was worn continuously throughout the intervention period, 24 hours a day. It was reapplied if participants reported detachment; otherwise, it was replaced every three days. In addition to taping, participants performed a corrective exercise program based on the NASM Corrective Exercise Continuum, which included four phases: inhibit, lengthen, activate, and integrate. The intervention lasted for three weeks, with 3 to 4 sessions per week, totaling 10 training sessions. Each session lasted approximately 60 to 75 minutes.
  Interventions: Device: Dynamic Tape; Device: Swiss Ball; Device: Dumbbells; Device: Visual Feedback Laser Device
- Dynamic Taping (DT Group) (Active Comparator): Participants in this group received postural taping using dynamic tape aimed at correcting forward head posture, rounded shoulders, and thoracic kyphosis. The taping method was identical to that used in the DT + EX group. The tape was worn continuously throughout the intervention period, 24 hours a day. It was reapplied if participants reported detachment; otherwise, it was replaced every three days. The intervention lasted for three weeks. No corrective exercise intervention was provided to this group.
  Interventions: Device: Dynamic Tape
- Corrective Exercise Group (EX Group) (Active Comparator): Participants in this group performed only the corrective exercise component used in the DT + EX group. The program was based on the NASM Corrective Exercise Continuum and included four phases: inhibit, lengthen, activate, and integrate. The intervention lasted for three weeks, with 3 to 4 sessions per week, totaling 10 training sessions. Each session lasted approximately 60 to 75 minutes. No taping was applied to this group.
  Interventions: Device: Swiss Ball; Device: Dumbbells; Device: Visual Feedback Laser Device
- Control Group (No Intervention): Participants in this group did not receive any intervention. They were instructed to maintain their usual daily activities and lifestyle throughout the three-week study period.

INTERVENTIONS:
Device: Dynamic Tape — Dynamic Tape is a viscoelastic tape designed to assist movement and absorb load. The material is composed of either Nylon/Lycra or Recycled PET/Lycra.
  Arms: Combined Dynamic Taping and Corrective Exercise (DT+EX Group); Dynamic Taping (DT Group)
Device: Swiss Ball — A 75 cm diameter Swiss ball was used to provide an unstable surface during the exercise intervention.
  Other Names: Therapy Ball
  Arms: Combined Dynamic Taping and Corrective Exercise (DT+EX Group); Corrective Exercise Group (EX Group)
Device: Dumbbells — During the exercise intervention, 1 kg and 2 kg dumbbells were used as external resistance.
  Arms: Combined Dynamic Taping and Corrective Exercise (DT+EX Group); Corrective Exercise Group (EX Group)
Device: Visual Feedback Laser Device — A headband was prepared to attach the laser pointer securely, allowing participants to wear it . This visual feedback laser device was used during proprioceptive training to provide real-time feedback.
  Arms: Combined Dynamic Taping and Corrective Exercise (DT+EX Group); Corrective Exercise Group (EX Group)

SUMMARY:
Upper Crossed Syndrome (UCS) is a pattern of muscle imbalance that leads to forward head posture, rounded shoulders, or excessive thoracic kyphosis, thereby affecting posture and cervical-shoulder function. Dynamic Taping is a taping technique aimed at enhancing movement control and muscle support through its elastic material and tension, influencing the skin and neuromuscular system. When applied to UCS patients, Dynamic Taping can assist in posture correction, improve posture control, and increase scapular dynamic stability. Additionally, Dynamic Taping can enhance proprioception, helping patients maintain proper posture through sensory feedback. Corrective exercises improve posture and stability by strengthening weakened muscles and stretching tight muscles. Combining these two interventions is expected to help address poor posture.

DETAILED DESCRIPTION:
This study aims to investigate the effects of Dynamic Taping combined with corrective exercises on cervical proprioception and muscle imbalance in UCS patients. A two-factor repeated measures ANOVA will be used to evaluate the effects before and after the intervention.

Participants recruited for this study must be adults aged 20 years or older. The study will evaluate their posture, including craniovertebral angle (CVA), sagittal shoulder angle (SSA), thoracic kyphosis angle, subacromial space, coracoid-humeral distance (CHD), cervical proprioception, muscle strength (deep cervical flexors, upper, middle, and lower trapezius, serratus anterior, rhomboid muscles), and electromyographic (EMG) to evaluate muscle activation (upper, middle, and lower trapezius, serratus anterior).

ELIGIBILITY:
Inclusion Criteria:

1. Age: >20years
2. Craniovertebral angle (CVA) of <48
3. Sagittal plane acromial angle of <52°
4. Thoracic kyphosis angle of >42° Meeting any one of these three angle conditions qualifies for inclusion.

Exclusion Criteria:

1. Allergic reactions to dynamic taping
2. Bodyweight outside the normal range (BMI between 18 and 25)
3. Any evident misalignment in the cervical spine, pelvis, or lower/upper limbs
4. Trunk rotation exceeding 5°during forward bending tests due to scoliosis
5. History of inherited muscle diseases, soft tissue lesions, or joint diseases involving the spine, scapulae, shoulders, abdomen, or pelvis
6. History of fractures or surgeries.
7. Inability to understand instructions

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Posture (CVA and SSA and Kyphosis Angle) | Participants were assessed at time points: prior to the intervention (baseline), immediately three weeks after the intervention, and at a one-month follow-up.
  The craniovertebral angle (CVA) and shoulder sagittal angle (SSA) were measured using the Physiomaster mobile application. During the measurement, the examiner positioned the smartphone to align the subject's image with the vertical and horizontal reference lines on the screen and then captured a photograph. The anatomical landmarks used for angle determination included the lateral canthus of the eye, the tragus of the ear, the spinous process of the seventh cervical vertebra (C7), and the midpoint of the line connecting the acromial processes.
  The thoracic kyphosis angle was measured using the Angle Meter mobile application. First, the device was calibrated to 0°. The smartphone was then placed at the level just inferior to T1 and subsequently at the level superior to T12. The kyphosis angle was calculated by summing the two measured angles.
Cervical Proprioception | Participants were assessed at time points: prior to the intervention (baseline), immediately three weeks after the intervention, and at a one-month follow-up.
  Cervical proprioception was assessed using the Head Repositioning Accuracy (HRA) test with a cervical range of motion (CROM) device. Participants were instructed to adopt and recognize the neutral head position (0°). The head was then passively guided to 30° of flexion, extension, lateral flexion, and rotation. After each movement, participants actively returned to the perceived neutral position under both eyes-open and eyes-closed conditions. The repositioning error was defined as the angular difference between the actual and the perceived 0° position

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy of China Medical University, Taichung, Beitun, Taiwan